CLINICAL TRIAL: NCT04848714
Title: Pharmacokinetic Study of ANAWIDOW [Antivenin Latrodectus (Black Widow) Equine Immune F(ab´)2] Solution 10 mL for Intravenous Use of Laboratorios Silanes, S.A. de C.V. in Healthy Adult Male and Female Subjects Under Fasting Conditions.
Brief Title: Pharmacokinetic Study Protocol of ANAWIDOW Lyophilized Powder for Solution for Intravenous Use in Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Collaborators: Rare Disease Therapeutics Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS/BW/ENE-21/0003
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Latrodectism
Keywords: Latrodectus envenomation; Black Widow; Equine immune; F(ab´)2
MeSH Terms: conditions — Spider Bites | interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group A: ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] (Experimental): ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] lyophilized powder for solution 10 mL
  Interventions: Drug: ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab)2] lyophilized powder for solution 10 mL

INTERVENTIONS:
Drug: ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab)2] lyophilized powder for solution 10 mL — Antivenin latrodectus (black widow) equine immune F(ab)2] lyophilized powder for solution 10 mL for intravenous use [parenteral formulation]; hence, a single-dose fasting pharmacokinetic study is planned.
  Other Names: ANAWIDOW

SUMMARY:
A single-dose, open-label, single-treatment, single-period pharmacokinetic study under fasting conditions, in 12 healthy adult. To evaluate the single dose pharmacokinetic profile ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] lyophilized powder for solution 10 mL (dose: 3x10 mL vials) for intravenous use.

DETAILED DESCRIPTION:
To evaluate the single dose pharmacokinetic profile ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] lyophilized powder for solution 10 mL (dose: 3x10 mL vials) for intravenous use of Laboratorios Silanes, S.A. de C.V. in healthy adult human male and female subjects under fasting conditions. To assess the safety of single dose of ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] lyophilized powder for solution 10 mL (dose: 3x10 mL vials) for intravenous use in healthy adult human male and female subjects under fasting conditions. In a minimum of 12 healthy adult. In this study, all subjects will be required to fast overnight for at least 10.00 hours prior to dosing at least 04.00 hours post-dose.

In this study, 3 ANAWIDOW 10 mL vials (3x10 mL) will be administered after diluting with normal saline solution up to 50 mL as intravenous infusion over 30 minutes. The solution will be infused through a 20-gauge catheter placed in the subject's left or right hand antecubital fossa at room temperature under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female subjects aged between 18 and 55 years (both inclusive).
* Subject is a light or non- or ex-smoker (A light smoker 1 being defined as someone who is smoking ≤ 9 cigarettes per day and an ex-smoker being defined as someone who completely stopped smoking for at least 6 months before screening): If any subject stops smoking during last 6 months before day of 1 of the study and smoke ≤ 9 cigarettes per day, the subject will also be considered as a light-smoker.
* With a weight ≥ 50.00 kg.
* With a body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 24.9 kg/m2.
* Found healthy according to the clinical laboratory results and physical examination (performed within 21 days prior to the dosing of the study).
* Have a normal 12-lead ECG and vital signs.
* Have laboratory test results within the laboratory's stated normal range, if not within this range, they must lack of clinical significance as judged by the PI or responsible physician.
* If the subject of the study is female and childbearing potential / fertile (a woman is considered fertile after menstruation and until she becomes postmenopausal, unless she is permanently sterile), and agrees to use ONE of the following methods during the study: 21 days before of the dosage and up to at least 28 days after the last administration of the study medication. 9. Women not considered of childbearing / fertile if they meet ONE of the following points:

  1. Postmenopausal for at least 1 year
  2. Premenopausal woman with ONE of the following:

     * hysterectomy
     * bilateral salpingectomy
     * bilateral oophorectomy
* The subject must be willing to use ONE of the following methods for 21 days before study drug dosing and at least 28 days after administration of the study medication;

  1. Willing to remain abstinent.
  2. Willing to use a male condom plus an additional contraceptive method.
* Be able to communicate effectively and voluntarily agreed to participate in this study by signing written informed consent after being informed sufficiently about study aspects like objectives, study procedures, characteristics of the investigational drug, expected adverse events.
* Subject willing to adhere to protocol requirements as evidenced by written informed consent approved by REC & RC.

Exclusion Criteria:

- Have any history of allergy or hypersensitivity to protein products of horse origin or IG or F(ab) or F(ab)2 or to any of its metabolites/derivatives or related drugs or excipients.

Or Study drug is contraindicated for medical reasons to the subject as per protocol section 3.7

* Have a positive test result for hepatitis B surface antigen (HBs Ag), hepatitis C virus antibody (HCV Ab), HIV antibodies (types 1 and 2) and/or VDRL.
* Have any history or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, hematological, dermatological, neurological or psychiatric disease or disorder (e.g., subjects with uncontrolled hypertension, phaeochromocytoma, carcinoid, thyrotoxicosis, bipolar depression, schizoaffective disorder and acute confusional states).
* Presence of gastrointestinal, hepatic or kidney disease, or surgery or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* Have a history of alcohol abuse or drug abuse.
* Have a history of smoking ≥ 10 cigarettes per day during the last 6 months prior to screening.
* History or presence of cancer.
* Have any history of gastrointestinal ulcers / intestinal bleeding.
* Have history of difficulty for donating blood.
* Have clinically significant abnormal laboratory tests results.
* Have a systolic blood pressure < 90 or > 140 mmHg or diastolic blood pressure is < 60 or > 90 mmHg.
* Have a pulse rate less than 60 bpm or greater than 100 bpm (lower range will be accepted up to 45 bpm in case of athlete).
* Have used any prescribed medication during the last 14 days preceding the first dosing, or use OTC, herbal products during the last 7 days or use medicinal enzyme inhibitors / inducers during las 30 days preceding the dosing.
* Have participated in a drug research study or donated blood within the last 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax). | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  To evaluate the single dose pharmacokinetic profile ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] lyophilized powder for solution 10 mL, employing the maximum observed concentration following the treatment (Cmax).
The area under the curve from time zero to the last measurable concentration (AUC 0-t)using the linear trapezoidal linear-interpolation method. | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  To evaluate the single dose pharmacokinetic profile ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] lyophilized powder for solution 10 mL, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t) using the linear trapezoidal linear-interpolation method.
The area under the curve from time zero to infinity calculated (AUC 0-inf). | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  The area under the curve from time zero to infinity calculated (AUC 0-inf). Where AUC0-inf = AUC0-t + Ct/ λz, Ct is the last measurable concentration, and λz is the terminal elimination rate constant.
Time of the maximum measured concentration (Tmax). | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  To evaluate the single dose pharmacokinetic profile ANAWIDOW [antivenin latrodectus (black widow) equine immune F(ab´)2] lyophilized powder for solution 10 mL, employing the time of the maximum measured concentration (Tmax).
First order rate constant associated with the terminal portion of the curve (log-lineal), Lambda_z (Kel). | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  This is estimated via linear regression of time vs log concentration data. This parameter will be calculated using at least three or more non-zero serum concentration values.
The elimination half-life (HL_Lambda_z (t½)) | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  The elimination half-life will be calculated as 0.693/ λz.
Vd (Volume of distribution) | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  A(t) (mg) / C(t) (mg/L) [A(t) represents the amount of drug in the body at time = t & C(t) represents serum / plasma concentration of the drug at time = t]
Clearance (CL) | Baseline, 00.08, 00.167, 00.25, 00.34, 00.50, 00.67, 00.83, 01.00, 01.50, 02.00, 04.00, 06.00, 12.00, 24.00,and 2, 3, 4, 6, 10, 14 and 21 days
  CL (body) = Kel x Vd (volume/hour)

SECONDARY OUTCOMES:
Physical examination | Baseline, 2, 3, 4, 6, 10, 14 and 21 days
  Physical examination will be performed before check-in of study period and may also be performed at any time during the study conduct if judged necessary by the physician.
Sitting blood pressure (mmHg) | Baseline, 2, 3, 4, 6, 10, 14 and 21 days
  Vital signs will be measured and registered at the time of check-in, prior to dosing, at 01.00, 03.00 and 05.00 hours (within a range of ± 45 minutes) after the same and before the check-out.
Pulse rate (p/m) | Baseline, 2, 3, 4, 6, 10, 14 and 21 days
  Vital signs will be measured and registered at the time of check-in, prior to dosing, at 01.00, 03.00 and 05.00 hours (within a range of ± 45 minutes) after the same and before the check-out.
Respiratory rate (rr) | Baseline, 2, 3, 4, 6, 10, 14 and 21 days
  Vital signs will be measured and registered at the time of check-in, prior to dosing, at 01.00, 03.00 and 05.00 hours (within a range of ± 45 minutes) after the same and before the check-out.
Axillary-body temperature (°C) | Baseline, 2, 3, 4, 6, 10, 14 and 21 days
  Vital signs will be measured and registered at the time of check-in, prior to dosing, at 01.00, 03.00 and 05.00 hours (within a range of ± 45 minutes) after the same and before the check-out.
Hematology & biochemistry laboratory tests | 21 days
  Hematology & biochemistry laboratory tests will be performed at the end of the study for all the subjects who administered with the study drug
Medical examination | Baseline, 2, 3, 4, 6, 10, 14 and 21 days
  It will be performed before check -in, prior to the dosing and before the check-out.
  Nevertheless, it may also be performed at any time during the study conduct if judged necessary by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Federico A Arguelles Tello, M.D, Principal Investigator — Avant Santé Research Center S.A. de C.V
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan NM, Buckley NA, Graudins A. Treatments for Latrodectism-A Systematic Review on Their Clinical Effectiveness. Toxins (Basel). 2017 Apr 21;9(4):148. doi: 10.3390/toxins9040148. PMID 28430165
- [Background] Vazquez H, Chavez-Haro A, Garcia-Ubbelohde W, Mancilla-Nava R, Paniagua-Solis J, Alagon A, Sevcik C. Pharmacokinetics of a F(ab')2 scorpion antivenom in healthy human volunteers. Toxicon. 2005 Dec 1;46(7):797-805. doi: 10.1016/j.toxicon.2005.08.010. Epub 2005 Sep 28. PMID 16197974
- [Background] Offerman SR, Daubert GP, Clark RF. The treatment of black widow spider envenomation with antivenin latrodectus mactans: a case series. Perm J. 2011 Summer;15(3):76-81. doi: 10.7812/TPP/10-136. PMID 22058673
- [Background] Dart RC, Bush SP, Heard K, Arnold TC, Sutter M, Campagne D, Holstege CP, Seifert SA, Lo JCY, Quan D, Borron S, Meurer DA, Burnham RI, McNally J, Garcia-Ubbelohde W, Anderson VE. The Efficacy of Antivenin Latrodectus (Black Widow) Equine Immune F(ab')2 Versus Placebo in the Treatment of Latrodectism: A Randomized, Double-Blind, Placebo-Controlled, Clinical Trial. Ann Emerg Med. 2019 Sep;74(3):439-449. doi: 10.1016/j.annemergmed.2019.02.007. Epub 2019 Mar 27. PMID 30926190
- See also: USFDA prescribing information ANAVIP® Crotalidae Immune F(ab')2 (Equine) Lyophilized Powder for Solution for Injection for Intravenous Use Only; Initial: 05/06/2015 — https://www.fda.gov/media/92139/download
- See also: Hilda Vázquez, Universidad Nacional Autónoma de México, Pharmacokinetics of a F(ab')(2) scorpion antivenom in healthy human volunteers — https://www.researchgate.net/publication/7567093_Pharmacokinetics_of_a_Fab_%272_scorpion_antivenom_in_healthy_human_volunteers
- See also: USFDA prescribing information ANASCORP® Centruroides (Scorpion) Immune F(ab')2 (Equine) Injection Lyophilized for Solution for intravenous use only; Revised: July 2011 — https://www.fda.gov/media/81093/download
- See also: Antivenin, black widow spider (Rx), Brand and Other Names: Antivenin (Latrodectus mactans), Medscape, Adverse Effects — https://reference.medscape.com/drug/latrodectus-mactans-antivenin-black-widow-spider-343717#4
- See also: A Phase III Multicenter Clinical Trial of Analatro® [Antivenin Latrodectus (Black Widow) Equine Immune F(ab)2] in Patients with Systemic Latrodectism; Instituto Bioclon S.A. de C.V — https://ichgcp.net/clinical-trials-registry/NCT00657540
- See also: USFDA. Retention of Bioavailability and Bioequivalence Testing Samples — https://www.fda.gov/ScienceResearch/SpecialTopics/RunningClinicalTrials/ucm120265.htm
- See also: Guideline for Good Clinical Practice, E6 (R2), International Council on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human use — https://www.fda.gov/media/93884/download